CLINICAL TRIAL: NCT03635164
Title: Phase I/Ib Trial of Radiotherapy in Combination With Durvalumab (MEDI4736) Prior to Surgical Resection for HPV Negative Squamous Cell Carcinoma of the Head and Neck (HNSCC)
Brief Title: Radiotherapy With Durvalumab Prior to Surgical Resection for HPV Negative Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-0606.cc
Record Dates: First submitted 2018-07-16; First posted 2018-08-17 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: HPV Negative; Durvalumab; Surgical Resection; Neoadjuvant; Radiation
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — durvalumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Expansion (Experimental): Part 1 of this trial will use a traditional 3+3 design will be used for this trial (i.e. cohort sizes of 3 patients for the first and second cohort at each dose level). Dose escalation will occur as long as there are minimal dose limiting toxicities.The expectation is that 9 patients will be enrolled to the trial during part 1.This is based on the expectation that all dose levels are safe (i.e. patients will not experience DLTs at all dose levels). The range of patients needed will be 6-12 patients.
  Part 2 of this trial will be an expansion cohort. A total of 8 additional patients will be enrolled at the dose level determined to be the MTD in part 1 of the study. These 8 patients will be used to confirm that the MTD is a safe combination, as well as provide additional patients to investigate the efficacy for the treatment combination.
  Note: Standard of care surgery will follow 3-6 weeks after medication and radiation treatment.
  Interventions: Drug: Durvalumab; Radiation: Stereotactic Body Radiation Therapy (SBRT); Procedure: Standard of Care Therapy

INTERVENTIONS:
Drug: Durvalumab — Patients will receive one dose of neoadjuvant durvalumab 1500 mg approximately 3-6 weeks prior to standard of care surgery. It will be given concurrently with the first dose of radiation (RT). Patients will receive up to six doses of durvalumab and radiation post-operatively.
Radiation: Stereotactic Body Radiation Therapy (SBRT) — The starting RT dose level will be given as 6 Gy for 2 fractions (12 Gy total) every other day over approximately one week to sites of gross disease only to minimize exposure to normal tissue. If toxicity develops and surgery is delayed by more than 8 weeks (qualifying as a DLT), the radiation dose will be dropped per protocol for the next set of patients. If this dose is tolerated, the dose will be increased to 6 Gy for 3 fractions (18 Gy total) for the next 3 patients.
Procedure: Standard of Care Therapy — Patients will proceed to surgical resection 3-6 weeks after radiation as recommended by the ENT surgeon.

SUMMARY:
This is a multi-center, prospective, single-arm phase I/Ib safety trial. Patients eligible for treatment must be diagnosed with non-metastatic, biopsy-proven stage II-IVB oral cavity, stage III-IVB larynx and hypopharynx, or stage III-IVB HPV/p16 negative intermediate-high risk oropharynx head and neck cancer, and must be eligible and amenable to surgical resection.

DETAILED DESCRIPTION:
This study will be enrolled using a 3+3 model. Patients will receive one dose of neoadjuvant durvalumab 1500 mg approximately 3-6 weeks prior to standard of care surgery. It will be given concurrently with the first dose of radiation (RT). The starting RT dose level will be given as 6 Gy for 2 fractions (12 Gy total) every other day over approximately one week to sites of gross disease (Table 1) only to minimize exposure to normal tissue. If toxicity develops and surgery is delayed by more than 8 weeks (qualifying as a DLT), the radiation dose will be dropped per protocol for the next set of patients. If this dose is tolerated, the dose will be increased to 6 Gy for 3 fractions (18 Gy total) for the next 3 patients. Patients will proceed to surgical resection approximately 3-6 weeks after radiation as recommended by the ENT surgeon.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed: stage II-IVB oral cavity, stage III-IVB larynx, stage III-IVB hypopharynx, or stage III-IVB HPV and/or p16 negative intermediate-high risk oropharynx head and neck cancer (AJCC 8th edition)
2. Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >10 mm by CT, PET/CT or MRI or >10 mm on visual inspection by clinical exam
3. Patients who are deemed resectable by ENT surgeon without pre-existing medical conditions that could inhibit surgery following neoadjuvant therapy, and do not refuse surgery
4. Written informed consent and HIPAA authorization obtained from the patient prior to performing any protocol-related procedures, including screening evaluations
5. Age > 18 years at time of study entry
6. ECOG performance status ≤ 1
7. Life expectancy ≥ 24 weeks
8. Body weight >30kg
9. Adequate normal organ and marrow function as defined below:

   * Hemoglobin ≥9.0 g/dL
   * Absolute neutrophil count (ANC) 1.0 x 109/L (> 1000 per mm3)
   * Platelet count ≥75 x 109/L (>75,000 per mm3)
   * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
   * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal
   * Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

Males:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

Females:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85

72 x serum creatinine (mg/dL)

10. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

* Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
* Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

  11. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 3 months
2. Patients with active ILD / pneumonitis or with a history of ILD/ pneumonitis requiring steroids
3. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
4. Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
5. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) 30 days prior to the first dose of study drug for patients who have received prior TKIs [e.g., erlotinib, gefitinib and crizotinib] and within 6 weeks for nitrosourea or mitomycin C. (If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period may be required.)
6. Patients with QTc interval > 470 msec during screening
7. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. The following are exceptions to this criterion:

   * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
   * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
   * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
8. Any concurrent chemotherapy, IP, biologic, or hormonal therapy that is not part of standard NCCN indicated HNSCC adjuvant concurrent CRT. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
9. History of allogenic organ or bone marrow transplantation
10. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    * Patients with celiac disease controlled by diet alone
11. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
12. History of another primary malignancy except for:

    * Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of IP and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
13. History of leptomeningeal carcinomatosis
14. History of active primary immunodeficiency
15. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
16. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
17. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ highly effective birth control from screening to 90 days after the last dose of durvalumab monotherapy. Patient must have a negative serum or urine pregnancy test within 72 hours of study entry.
18. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
19. Prior randomisation or treatment in a previous durvalumab clinical study
20. Patients with p16-positive oropharyngeal SCCA. No verification of p16 status is needed for laryngeal cancer or oral cavity cancer.
21. Patients with sinonasal SCCAs
22. Patients with metastatic SCCA neck disease with an unknown primary tumor site
23. Patients with distant metastatic disease on initial screening imaging
24. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose and Dose Limiting Toxicities | Study start date to study end date, or death, whichever comes first, up to 24 months
  The Maximum Tolerated Dose (MTD) and Dose Limiting Toxicities (DLT) will be discovered by using the 3+3 study design.

SECONDARY OUTCOMES:
Pathologic Response | Study start date to study end date, or death, whichever comes first, up to 24 months
  Tumor response to neoadjuvant therapy (durvalumab + SBRT) will be assessed by pathology review of the surgical specimen. Response will be labeled as complete pathologic remission, microscopic residual tumor (only scattered foci of residual tumor cells) or macroscopic residual tumor.
Clinical Response | Study start date to study end date, or death, whichever comes first, up to 24 months
  Overall survival (OS), along with locoregional control and distant control will be determined from the time of enrollment to date of death due to any cause. OS will be evaluated by Kaplan-Meier estimate.
Evaluate Biomarkers: Gene Expression | Study start date to study end date, or death, whichever comes first, up to 24 months
  Analysis of gene expression of RNA levels and entire genome sequences using the 10X Genomics single-cell RNA-sequencing platform.
Evaluate Biomarkers: Phenotypic Analysis | Study start date to study end date, or death, whichever comes first, up to 24 months
  Phenotypic analysis of T cells and assessment of intracellular and circulating cytokines using multiplex mass flow cytometry to analyze phenotypic changes, functional response of cytokine production, and activation status of tumor infiltrating lymphocytes (TILs), circulating T cells (especially CD8 and PD-1 expression), and peripheral blood mononuclear cells (PBMCs).
Evaluate Biomarkers: Immune Cell Infiltration | Study start date to study end date, or death, whichever comes first, up to 24 months
  Examination of intratumoral immune cell infiltration using the Perkin Elmer Vectra 3 and tissue microarrays.
Toxicity Profile | Study start date to study end date, or death, whichever comes first, up to 24 months
  Grading of adverse effects (AEs) will follow the guidelines provided in the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Short Term Quality of Life | Study start date to study end date, or death, whichever comes first, up to 24 months
  Short- and long-term quality of life will be obtained using FACT H&N v4 and will be assessed at baseline, with each cycle, post-SBRT, post-surgically, and throughout adjuvant therapy on a standard schedule.

CONTACTS AND LOCATIONS:
Overall Officials: Sana Karam, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University of Colorado Hospital, Aurora, Colorado
  - Memorial Hospital Central, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado

REFERENCES:
- [Derived] Darragh LB, Knitz MM, Hu J, Clambey ET, Backus J, Dumit A, Samedi V, Bubak A, Greene C, Waxweiler T, Mehrotra S, Bhatia S, Gadwa J, Bickett T, Piper M, Fakhoury K, Liu A, Petit J, Bowles D, Thaker A, Atiyeh K, Goddard J, Hoyer R, Van Bokhoven A, Jordan K, Jimeno A, D'Alessandro A, Raben D, McDermott JD, Karam SD. A phase I/Ib trial and biological correlate analysis of neoadjuvant SBRT with single-dose durvalumab in HPV-unrelated locally advanced HNSCC. Nat Cancer. 2022 Nov;3(11):1300-1317. doi: 10.1038/s43018-022-00450-6. Epub 2022 Nov 25. PMID 36434392